CLINICAL TRIAL: NCT03529097
Title: Randomized Controlled Trial to Evaluate the Efficiency of IV Fluids in the Treatment of Renal Colic
Brief Title: Evaluation of the Roll of IV Fluids in the Treatment of Renal Colic
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolles
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-18-4262-NK-CTIL
Record Dates: First submitted 2018-04-23; First posted 2018-05-18 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2018-04

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Sodium Chloride; Dipyrone; Diclofenac; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluids (Active Comparator): Intervention: 2 liters of 0.9% NaCl IV during the ER stay with pain killers. For placebo purposes this arm participants will get an infusion with black cover so they could not tell if it drips or not
  Interventions: Drug: 0.9% Sodium-chloride; Drug: Optalgin, Voltaren, Morphine
- Placebo (Placebo Comparator): No interventions, Only pain killers. For placebo purposes this arm participants will get an infusion with black cover so they could not tell if it drips or not
  Interventions: Drug: Placebos; Drug: Optalgin, Voltaren, Morphine

INTERVENTIONS:
Drug: 0.9% Sodium-chloride — 2 liters of 0.9% NaCl IV fluids
  Arms: Fluids
Drug: Placebos — 2 liters of 0.9% NaCl bag covered with black bag so the participant could not tell the fluids are not dripping to his vain
  Arms: Placebo
Drug: Optalgin, Voltaren, Morphine — Oral and IV Optalgin, Voltaren IM (intramuscular), Morphine IV. All according to the pain intensity and with concordance to the physician.

SUMMARY:
A randomised controlled trial to evaluate the role of IV fluids in renal colic.

DETAILED DESCRIPTION:
A RCT (Randomized Controlled Trial)to evaluate the role of 0.9% NACL (sodium chloride) IV fluids during an acute renal colic. The 2 arms will include -

1. 2 liters of 0.9% NACL IV fluids with pain killers
2. only pain killers The object is to find out if the IV fluids has any advantage in the care of renal colic. Does it helps to relive the pain? Does the stone eject earlier? Will there be fewer interventions?

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* clinical renal colic
* a radiological proof (CT,US) to urolithiasis

Exclusion Criteria:

* below 18 years
* has a contraindication for IV fluids (such as CHF (Congestive Heart Failure)etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone ejection without intervention | 1 month
  Has the stone ejected without intervention? 1 month after the first visit in the ER (Emergency Room) we will preform an US or CT exam to verified that the stone ejected. If the stone that was seen by the US or CT in the ER is not present after 1 month we will assume it was spontaneously ejected. we would like to find out if there is any differences between the 2 groups in matter of spontaneously stone ejection. (Yes or No)
The need for urological intervention | 0 to 1 month
  The need for urological intervention. 1 month after the visit in the ER we will check if the patient have gone through urological intervention such as urolithiasis. We would like to find out if there is any difference between the two groups in matter of urological intervention between 1 month after the visit in the ER. (Yes or No)
Pain | 6 hours
  Measure the VAS (Visual Analogue pain Score). Between 1-10 1 is no pain and 10 in the strongest pain. a scale between 1-10 is shown to the patients and they are asked how they feel after 6 hours of treatment in the ER

SECONDARY OUTCOMES:
Pain | 1 Hour
  Measure the VAS Between 1-10 1 is no pain and 10 in the strongest pain. a scale between 1-10 is shown to the patients and they are asked how they feel after 1 hour of treatment in the ER
Pain | 1 month
  Measure the VAS Between 1-10 1 is no pain and 10 in the strongest pain. a scale between 1-10 is shown to the patients and they are asked how they feel after 1 month from the first visit in the ER

IPD SHARING:
Plan to Share IPD: No